CLINICAL TRIAL: NCT02361047
Title: Healthy Kids After Cancer: A Physical Activity and Nutrition Intervention
Brief Title: Let's Play! Healthy Kids After Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Masonic Cancer Center, University of Minnesota (Other); Children's Hospitals and Clinics of Minnesota (Other); St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A13-175; 1R21CA182727-01A1 (NIH)
Record Dates: First submitted 2015-01-23; First posted 2015-02-11 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Childhood Acute Lymphoblastic Leukemia in Remission; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phone Coaching Program (Experimental): Participants will receive a nutrition and physical activity phone coaching program, in addition to standard-of-care physician counseling regarding lifestyle recommendations to achieve/maintain a healthy weight trajectory after cancer treatment.
  Interventions: Behavioral: Phone Coaching Program
- Standard Care Control (No Intervention): Participants will receive standard-of-care physician counseling regarding lifestyle recommendations to achieve/maintain a healthy weight trajectory after cancer treatment.

INTERVENTIONS:
Behavioral: Phone Coaching Program — Participants in this group will receive a 10-session nutrition and physical activity program delivered via phone by a health behavior coach to promote healthy lifestyle changes. Participants will also receive standard-of-care physician counseling regarding lifestyle recommendations to achieve/maintain a healthy weight trajectory after cancer treatment.
  Arms: Phone Coaching Program

SUMMARY:
This pilot study will evaluate the feasibility, acceptability, and potential efficacy of a parent-targeted, phone-based program to prevent unhealthy weight gain and improve biomarkers of oxidative stress and inflammation among childhood acute lymphoblastic leukemia survivors.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is the most common childhood cancer, accounting for 25% of all childhood malignancies. Treatment of childhood ALL has a high success rate, with long-term event-free survival of >85%. Treatment success, however, has not come without cost. Recognition of long-term health problems related to childhood cancer therapies is growing. Both during and after therapy, children treated for ALL are at risk for fatigue, reduced physical activity, poor dietary intake, and excessive weight gain, which are driven by physiological (chemotherapy-induced) changes and social (home/environmental) factors. The goals of this pilot study are to evaluate the feasibility, acceptability, and potential efficacy of a parent-targeted, phone-delivered nutrition and physical activity program to prevent unhealthy weight gain among 60 childhood ALL survivors, 4-10 years of age. Participants will be randomly assigned to either the phone-delivered parent-targeted nutrition and physical activity intervention or a standard-of-care control group. Intervention success will be benchmarked by changes in key weight-related behaviors (physical activity and dietary intake) over the 6-month trial, and initial impact of the intervention on biomarkers of inflammation and oxidative stress, fatigue, and body composition will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Between 4.0 years and < 11.0 years of age at the time of recruitment
* Previously diagnosed of ALL and currently in remission
* Between 1-5 years post completion of chemotherapy
* BMI ≥ 85 percentile for age and sex (overweight or obese) OR at risk for obesity (BMI between the 50th and 85th percentile and at least one overweight parent (BMI ≥ 25 kg/m2)

Exclusion Criteria:

* History of cranial radiation therapy
* History of bone marrow transplant
* History of relapse of ALL
* Diagnosis of Down's Syndrome
* Comorbidities of obesity that require immediate subspecialist referral
* Significant pulmonary, cardiovascular, orthopedic, or musculoskeletal problems that would, in their oncologist's judgment, limit their ability to participate in physical activity
* Significant psychiatric or neurologic disorders that would impair compliance with study protocol
* Current participation in a weight-loss program

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Feasibility: Number of participants who complete 8 of 10 intervention sessions | 6 months
  Measured by intervention session completion rates.
Retention: Number of participants who complete 6-month outcome assessments | 6 months
  Measured by completion of the 6-month outcome assessment.
Acceptability: Number of participants who report high satisfaction with the intervention | 6 months
  Measured by parent survey of satisfaction with intervention materials and sessions.

SECONDARY OUTCOMES:
Change in children's physical activity | 6 months
  Measured by ActiGraph accelerometers
Change in children's dietary intake | 6 months
  Measured by Nutrition Data System for Research (NDSR) interview
Change in children's BMI | 6 months
  Staff-measured height and weight
Change in children's biomarker outcome measures | 6 months
  Measured by serum blood samples
Change in children's energy level | 6 months
  Measured by questionnaire: PedsQL Multidimensional Fatigue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alicia S Kunin-Batson, PhD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Background] Rogers PC, Meacham LR, Oeffinger KC, Henry DW, Lange BJ. Obesity in pediatric oncology. Pediatr Blood Cancer. 2005 Dec;45(7):881-91. doi: 10.1002/pbc.20451. PMID 16035086
- [Background] Ness KK, Armenian SH, Kadan-Lottick N, Gurney JG. Adverse effects of treatment in childhood acute lymphoblastic leukemia: general overview and implications for long-term cardiac health. Expert Rev Hematol. 2011 Apr;4(2):185-97. doi: 10.1586/ehm.11.8. PMID 21495928
- [Background] Ness KK, Leisenring WM, Huang S, Hudson MM, Gurney JG, Whelan K, Hobbie WL, Armstrong GT, Robison LL, Oeffinger KC. Predictors of inactive lifestyle among adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Cancer. 2009 May 1;115(9):1984-94. doi: 10.1002/cncr.24209. PMID 19224548
- [Background] Cohen J, Wakefield CE, Fleming CA, Gawthorne R, Tapsell LC, Cohn RJ. Dietary intake after treatment in child cancer survivors. Pediatr Blood Cancer. 2012 May;58(5):752-7. doi: 10.1002/pbc.23280. Epub 2011 Aug 17. PMID 21850679
- [Background] Mayer EI, Reuter M, Dopfer RE, Ranke MB. Energy expenditure, energy intake and prevalence of obesity after therapy for acute lymphoblastic leukemia during childhood. Horm Res. 2000;53(4):193-9. doi: 10.1159/000023566. PMID 11044803
- [Background] Sherwood NE, Levy RL, Langer SL, Senso MM, Crain AL, Hayes MG, Anderson JD, Seburg EM, Jeffery RW. Healthy Homes/Healthy Kids: a randomized trial of a pediatric primary care-based obesity prevention intervention for at-risk 5-10 year olds. Contemp Clin Trials. 2013 Sep;36(1):228-43. doi: 10.1016/j.cct.2013.06.017. Epub 2013 Jun 28. PMID 23816490